CLINICAL TRIAL: NCT06121596
Title: Relaxation Effects of Personalized Breathing Exercises for Healthy College Students: a Randomized Crossover Trial
Brief Title: Relaxation Effects of Personalized Breathing Exercises for Healthy College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Lukas Moebus, Principal Investigator, Technical University of Munich
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: P-BP-40-60-80-RCT
Record Dates: First submitted 2023-08-10; First posted 2023-11-08 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Breathing Exercises
Keywords: Relaxation therapy; Stress-management; Breathing exercise; Stress; Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Breathing Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Breathing Exercise with 40 Percent of the Spontaneous Breathing Frequency (A) (Experimental): Participants are instructed (via visual pacer) to reduce their breathing frequency to 40 percent of their spontaneous breathing frequency for a period of five minutes. In advance, participants are instructed (via pre-recorded video) to breathe nasally (if possible) and abdominally, with a prolonged exhalation (inspiration-to-expiration ratio is 1-to-2 - also instructed via visual pacer) during the breathing exercise.
  Interventions: Behavioral: Breathing Exercise
- Breathing Exercise with 60 Percent of the Spontaneous Breathing Frequency (B) (Experimental): Participants are instructed (via visual pacer) to reduce their breathing frequency to 60 percent of their spontaneous breathing frequency for a period of five minutes. In advance, participants are instructed (via pre-recorded video) to breathe nasally (if possible) and abdominally, with a prolonged exhalation (inspiration-to-expiration ratio is 1-to-2 - also instructed via visual pacer) during the breathing exercise.
  Interventions: Behavioral: Breathing Exercise
- Breathing Exercise with 80 Percent of the Spontaneous Breathing Frequency (C) (Experimental): Participants are instructed (via visual pacer) to reduce their breathing frequency to 80 percent of their spontaneous breathing frequency for a period of five minutes. In advance, participants are instructed (via pre-recorded video) to breathe nasally (if possible) and abdominally, with a prolonged exhalation (inspiration-to-expiration ratio is 1-to-2 - also instructed via visual pacer) during the breathing exercise.
  Interventions: Behavioral: Breathing Exercise

INTERVENTIONS:
Behavioral: Breathing Exercise — A breathing exercise is a relaxation technique (or therapy) to increase relaxation (induces a relaxation response) and decrease stress (reduces a stress response).

SUMMARY:
Stress plays a major role in the etiology and pathogenesis of anxiety and depression. Relaxation therapies, such as breathing exercises, can reduce stress and increase relaxation.

This study has two aims. First, it aims to personalize and optimize breathing protocols. Second, it aims to tailor breathing protocols to subgroups based on prediction models of expected efficacy.

Three different breathing protocols, varying solely in their instructed breathing frequency with 40 percent (A), 60 percent (B), and 80 percent (C) of the interindividual spontaneous breathing frequency, are tested in a randomized, counterbalanced crossover trial. Other parameters, such as breathing quality (i.e., nasal and diaphragmatic), rhythm (i.e., prolonged exhalation without instructed pauses) and depth (i.e., increased depth due to slower breathing frequency) as well as contextual factors (e.g., posture, video-based instructions, type of pacer, etc.) are invariant between protocols.

First, this study hypothesizes a difference in the relaxation response between breathing protocols A, B, and C. This study looks at the relaxation response from three different angles (1) self-report, (2) autonomic arousal, and (3) central nervous system arousal. Second, this study explores prediction models of expected efficacy based on the interindividual variance in characteristics (i.e., depressive, anxious and stress symptoms as well as expertise in relaxation therapies) and biomarkers (e.g., heart rate variability, peripheral temperature, skin conductance, etc.). Prediction models can tailor breathing protocols to subgroups to increase expected efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years old
* University student
* Native German speaker

Exclusion Criteria:

* Any psychiatric (e.g., anxiety), neurologic (e.g., epilepsy) or cardio-pulmonary (e.g., asthma) diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Relaxation Sum Score | Immediately after each 5-minute breathing exercise
  Measured with the German Version of the Relaxation State Questionnaire; Sum scores range from 10 to 50 (higher scores indicate greater relaxation).

SECONDARY OUTCOMES:
Current Perceived Stress Level | Immediately after each 5-minute breathing exercise
  Measured on a visual analog scale ranging from 0 to 100, where zero is absolutely no stress and 100 is extreme stress.
Heart Rate Variability | During each 5-minute breathing exercise
  Measured via blood volume pulse with a finger clip on the middle finger
Peripheral Temperature | During each 5-minute breathing exercise
  Measured via temperature sensor on the small finger
Skin Conductance | During each 5-minute breathing exercise
  Measured via skin conductance sensor on the index and ring finger
Power in Frequency Bands | During each 5-minute breathing exercise
  Measured via four channel EEG with linked earlobe reference and active electrode placement on F3, F4, F7, and F8 according to the international 10-20 system

OTHER OUTCOMES:
Breathing Frequency | During the first questionnaire and video-based instructions before the baseline measurement, the 5-minute baseline measurement and during each 5-minute breathing exercise
  Measured via chest strap sensor. This is not an outcome, it measures the participant's spontaneous breathing frequency and the compliance to the breathing protocols.
Number of Participants with Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | Immidiately after the last breathing exercise
  Assessed with a questionnaire. This is not an outcome measure, this is a measure to build a prediction model for expected efficacy of breathing exercises.
Difficulty with any of the Breathing Exercises | Immidiately after the last breathing exercise
  Assessed with a questionnaire. This is not an outcome measure, this is a measure to build a prediction model for expected efficacy of breathing exercises.
Transferability of Breathing Exercises into Daily Life | Immidiately after the last breathing exercise
  Assessed with a questionnaire. This is not an outcome measure, this is a measure to build a prediction model for expected efficacy of breathing exercises.
One Word Description for Breathing Exercises | Immidiately after the last breathing exercise
  Assessed with an open question. This is not an outcome measure, this is a measure to build a prediction model for expected efficacy of breathing exercises.
Previous Training in Relaxation Techniques (such as Breathing Exercises, Autogenic Training, Progressive Relaxation, etc.) | Immidiately after the last breathing exercise
  Assessed with a closed (Yes/No) question. This is not an outcome measure, this is a measure to build a prediction model for expected efficacy of breathing exercises.
Duration of Training in Relaxation Techniques (such as Breathing Exercises, Autogenic Training, Progressive Relaxation, etc.) | Immidiately after the last breathing exercise
  Assessed with a questionnaire. This is not an outcome measure, this is a measure to build a prediction model for expected efficacy of breathing exercises.
Average Volume of Training in Relaxation Techniques (such as Breathing Exercises, Autogenic Training, Progressive Relaxation, etc.) | Immidiately after the last breathing exercise
  Assessed with a questionnaire. This is not an outcome measure, this is a measure to build a prediction model for expected efficacy of breathing exercises.
Stress, Anxiety and Depression Score of the Past Two Weeks | Immidiately after the last breathing exercise
  Measured with the Depression-Anxiety-Stress-Scale Questionnaire. This is not an outcome measure, this is a measure to build a prediction model for expected efficacy of breathing exercises.

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Moebus, M.Sc., Principal Investigator — Technical University of Munich
Locations (1):
- Technical University of Munich, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Yes